CLINICAL TRIAL: NCT00033566
Title: A Phase I Study of S-3304 in Patients With Solid Tumors
Brief Title: S-3304 in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Patrick Creaven, MD, Roswell Park Cancer Institute
Purpose: Treatment
Other Study IDs: CDR0000069301; RPCI-DS-0120
Record Dates: First submitted 2002-04-09; First posted 2003-01-27 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — S 3304

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: S-3304

SUMMARY:
RATIONALE: S-3304 may stop or slow the growth of solid tumors by stopping blood flow to the tumor.

PURPOSE: Phase I trial to study the effectiveness of S-3304 in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and safety profile of S-3304 in patients with advanced solid tumors.
* Determine the pharmacokinetic profile of this drug in these patients.
* Estimate the starting dose of this drug for subsequent phase II efficacy studies.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral S-3304 twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 6-8 patients receive escalating doses of S-3304 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 or 3 of 8 patients experience dose-limiting toxicity.

Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 6-28 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor that failed to respond or relapsed after prior therapy or for which no standard therapy exists
* Biopsy-accessible lesion
* No brain metastasis unless clinically stable and off therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 6 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* Transaminases less than 2.5 times ULN

Renal:

* Creatinine less than 2.0 mg/dL

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 30 days after study
* Able to tolerate oral medication
* HIV negative
* No AIDS
* No serious underlying gastrointestinal disorders (e.g., recurrent vomiting or inflammatory bowel disease)
* No other serious concurrent illness

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy
* Concurrent stable doses of epoetin alfa are allowed during the second and subsequent courses
* No other concurrent immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since prior hormonal therapy
* Concurrent stable doses of steroids for prostate cancer are allowed during the second and subsequent courses
* No concurrent hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* No prior significant gastric resection

Other:

* Recovered from prior therapy
* At least 4 weeks since other prior investigational antitumor drugs
* No other concurrent investigational antitumor drugs
* Concurrent stable doses of bisphosphonates, cyclo-oxygenase-2 inhibitors, and non-steroidal anti-inflammatory drugs are allowed during the second and subsequent study courses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2002-12 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Creaven, MBBS, PhD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] Chiappori AA, Eckhardt SG, Bukowski R, Sullivan DM, Ikeda M, Yano Y, Yamada-Sawada T, Kambayashi Y, Tanaka K, Javle MM, Mekhail T, O'bryant CL, Creaven PJ. A phase I pharmacokinetic and pharmacodynamic study of s-3304, a novel matrix metalloproteinase inhibitor, in patients with advanced and refractory solid tumors. Clin Cancer Res. 2007 Apr 1;13(7):2091-9. doi: 10.1158/1078-0432.CCR-06-1586. PMID 17404091